CLINICAL TRIAL: NCT02449954
Title: Comparison Between the Effects of Intravenous Morphine, Tramadol and Ketorolac on Stress and Immune Responses in Patients Undergoing Modified Radical Mastectomy
Brief Title: Effect of Morphine, Tramadol, and Ketorolac on Postoperative Stress and Immune Responses
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmad Mohammad Abd El-Rahman, Lecturer, Assiut University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 43
Record Dates: First submitted 2015-04-29; First posted 2015-05-21 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Breast Cancer
Keywords: Stress and Immune Responses; morphine; tramadol; ketorolac
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- morphine group (Active Comparator): intravenous 0.1mg/kg morphine
  Interventions: Drug: Intravenous morphine sulphate
- tramadol group (Active Comparator): intravenous 2 mg/kg tramadol
  Interventions: Drug: Intravenous tramadol HCL
- ketorolac group (Active Comparator): intravenous30 mg ketorolac
  Interventions: Drug: Intravenous ketorolac tromethamine

INTERVENTIONS:
Drug: Intravenous morphine sulphate — Group I:received IV 0.1mg/kg morphine sulphate.
  Other Names: venous blood samples
  Arms: morphine group
Drug: Intravenous tramadol HCL — Group II:received IV 2 mg/kg tramadol HCL.
  Other Names: venous blood samples
  Arms: tramadol group
Drug: Intravenous ketorolac tromethamine — Group III: received IV 30 mg ketorolac tromethamine
  Other Names: venous blood samples
  Arms: ketorolac group

SUMMARY:
Comparison between the effects of intravenous morphine, tramadol and ketorolac on stress and immune responses in patients undergoing modified radical mastectomy

DETAILED DESCRIPTION:
Sixty patients aged (20-60 years), weighting (50 -75 Kg), with American Society of Anesthesiologists (ASA) physical status I or II scheduled for modified radical mastectomy surgery under general anesthesia were enrolled in this prospective clinical study. The Ethics Committee of South Egypt Cancer Institute (SECI), assuit University, assuit, Egypt approved the study. Informed written consent was obtained from each patient to be enrolled in this study.

Patients with known allergy to opioids or Non Steroidal Anti-inflammatory drugs NSAIDs, with gastric or duodenal ulcer, on radiotherapy or chemotherapy, received blood transfusion before the surgery or preoperative NSAIDs, steroid or opioid medications 48 hours prior to operation were excluded.

All patients were taught how to evaluate their own pain intensity using the visual analogue scale (VAS) scored from 0 to 10 (where 0 = no pain and 10 = the worst pain imaginable). Both the patient and the anesthetist involved in the study were kept blinded to group assignment. Randomization codes were not decoded till the end.

No pre-medications were given. Basic monitoring probes (ECG, non invasive blood pressure, end-tidal carbon dioxide, pulse oximetry and temperature) were applied. base line VAS, sedation score, systolic and diastolic blood pressure, heart rate, respiratory rate and oxygen saturation were assessed before the beginning of surgery. Venous blood sample was taken for assessment of the base line stress hormones (cortisol, prolactin) and immune response (cluster of differentiation (CD) 3, 4, 8 and 56), General anesthesia was induced with I.V. fentanyl 1 μg/kg, thiopental 5mg/kg. Endotracheal intubation was facilitated by cis-atracurium 0.15 mg/kg, and was maintained with isoflurane 1.5-1.7 MAC, cis-atracurium 0.03 mg/kg and controlled ventilation in a ventilation parameters that maintain normocapnia (35- 45 mmHg). Neuromuscular block was antagonized by neostigmine 50µg/kg and atropine 20µg/kg. Venous blood sample was taken for assessment of stress hormones (cortisol, prolactin) and immune response (CD3, CD4, CD8 and CD56) immediately postoperatively after extubation in the operative room before the analgesic drug administration. VAS, sedation score, systolic and diastolic blood pressure, heart rate, respiratory rate and oxygen saturation were also assessed. Patients were allocated according to computer-generated randomization tables into one of three groups of 20 patients each to receive:

Group I: (n=20) received IV 0.1mg/kg morphine sulphate (morphine sulfate ®, Misr CO Pharma).

Group II: (n=20) received IV 2 mg/kg tramadol Hcl (tramadol ®, October Pharma S.A.E).

Group III: (n=20) received IV 30 mg ketorolac tromethamine (ketorolac ®, Amriya Pharma).

Patients were transferred to the post anesthesia care unit (PACU). During this period observation of heart rate, systolic and, diastolic blood pressure, respiratory rate, oxygen saturation and VAS were recorded at 2, 4, 6, 8, 12, 18 and 24hrs postoperatively. In addition, side effect such as nausea, vomiting, respiratory depression and sedation (using sedation score from 0 to 4, where 0= awake, 1= easily aroused, 2= awaken after verbal stimulation, 3=awaken after tactile stimulation and 4= not arousable) were recorded and treated. Another venous blood samples were taken for assessment of stress hormones at 40 mins, immune response at 90 mins and for both stress hormones and immune responses at 24 hours later. In order to keep VAS ≤ 3 for 24hours postoperative, repeated doses of the same analgesic medications (morphine to the first group, tramadol to the second group, and ketorolac to the third group) were given all over the observation period at the same doses.

Determination of serum cortisol and prolactin levels was done by fully automated ELISA (enzyme linked immunosorbent assay) (EVOLIS®, Biorad, Germany). Expressions of (CD3+, CD4+, CD8+ and CD56+) in blood samples were measured as percentages of total lymphocytes by fluorescence activated cell sorter (FACS) calibur flow cytometry with cell quest software (Becton Dickinson Biosciences, USA). Anti-human IgG was used as an iso type-matched negative control for each sample. Forward and side scatter histogram was used to define the lymphocyte population. Then, the percentages of CD3+, CD4+, CD8+ and CD56 were assessed in lymphocytes population. The positive percentage was >20%

ELIGIBILITY:
Inclusion Criteria:

* patients aged (20-60 years)
* weighting (50 -75 Kg),
* with American Society of Anesthesiologists (ASA) physical status I or II

Exclusion Criteria:

* Patients with known allergy to opioids or NSAIDS,
* gastric or duodenal ulcer, on radiotherapy or chemotherapy
* received blood transfusion before the surgery or preoperative NSAIDs, steroid or opioid medications 48 hours prior to operation

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-06; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Serum cortisol level | 11 month
  was measure by fully automated ELISA
Serum prolactin level | 11 month
  was measure by fully automated ELISA
Expression of peripheral T lymphocytes subset cluster of differentiation3 percentage(CD3+) | 11 month
  was measured by flow cytometry
Expression of peripheral T lymphocytes subset cluster of differentiation 4 percentage (CD4+) | 11 month
  was measured by flow cytometry
Expression of peripheral T lymphocytes subset cluster of differentiation 8 percentage (CD8+) | 11 month
  was measured by flow cytometry
Expressions of peripheral T lymphocytes subset cluster of differentiation56 percentage (CD56+) | 11 month
  was measured by flow cytometry